CLINICAL TRIAL: NCT06247033
Title: Evaluation of the Efficacy of Transcutaneous Tibial Nerve Stimulation on Post-Stroke Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Umay Ekinci, MD, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 42
Record Dates: First submitted 2024-01-21; First posted 2024-02-07 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-01

CONDITIONS: Incontinence, Urge; Stroke; Neurogenic Bladder
MeSH Terms: conditions — Urinary Incontinence, Urge; Stroke; Urinary Bladder, Neurogenic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active TNS - Chronic stroke patients with urgency symptoms, followed with PFTE, BT, TNS (Active Comparator): Study group was followed with tibial nerve stimulation for 6 weeks, 2 sessions in a week, for 30 minutes. Stimulation was performed with TENS device, with settings of 10 Hz frequency, 200 msn wavelenght, continuous symetrical biphasic current. Amptlitude was increased just below the motor range that cause flexion in toes. All patiens were followed for PFTE and BT according to standard schedule.
  Interventions: Device: Tibial Nerve Stimulation with TENS device
- Sham TNS - Chronic stroke patients with urgency symptoms, followed with PFTE, BT, Sham TNS (Sham Comparator): Control group was followed with sham tibial nerve stimulation, which were performed by after starting electric current with TENS device, current were decreased and completely shut down. Sham stimulation was also applied for 6 weeks, 2 times in a week, 30 minutes. All patients were followed for PFTE and BT according to given standard schedule.
  Interventions: Behavioral: Pelvic muscle training exercise with bladder training

INTERVENTIONS:
Device: Tibial Nerve Stimulation with TENS device — Tibial nerve stimulation was applied with TENS device transcutaneously and electrodes were positioned in medial part of the ankle. Negative transcutaneous electrode was positioned 3 centimeter posteriorly to the medial malleol. And positive transcutaneous electrode was positioned 10 centimeter above the negative electrode.
  Arms: Active TNS - Chronic stroke patients with urgency symptoms, followed with PFTE, BT, TNS
Behavioral: Pelvic muscle training exercise with bladder training — Control group was followed with sham tibial nerve stimulation, which were performed by after starting electric current with TENS device, current were decreased and completely shut off. Sham stimulation was also applied for 6 weeks, 2 times in a week, 30 minutes. All patients were followed for PFTE and BT according to given standard schedule.
  Arms: Sham TNS - Chronic stroke patients with urgency symptoms, followed with PFTE, BT, Sham TNS

SUMMARY:
The goal of this clinical trial is to comparing the efficacies of different managements in patients with overactive bladder symptoms with stroke

The main question it aims to answer are:

* Are pelvic floor training exercises and bladder training enough to ease the symptoms of overactive bladder in patients with stroke?
* Is tibial nerve stimulation really effective and does it decrease the need of medications in patients with overactive bladder with stroke? Participants are questioned if they have the symptoms of overactive bladder. After urodynamic evaluation, they are separated in 2 groups. Pelvic floor training exercises and bladder training are given in both groups; while one of the groups is followed with tibial nerve stimulation and the other one is followed with sham tibial nerve stimulation for 6 weeks.

Our main aim was to compare effectiveness of tibial nerve stimulation in patiens with overactive bladder with stroke.

DETAILED DESCRIPTION:
A sham-controlled double-blinded randomized study was undertaken. 28 patients with chronic stroke were randomized into 2 groups. Pelvic floor training exercises and bladder training are given in both groups; while one of the groups is followed with tibial nerve stimulation and the other one is followed with sham tibial nerve stimulation for 6 weeks.

In both groups, patients are followed for completing the standart schedule of PFTE and BT; and excluded from our study if their rates below %80 according to exercise and training schedule.

Study group was followed with tibial nerve stimulation for 6 weeks, 2 sessions in a week, for 30 minutes. Stimulation was performed with TENS device, with settings of 10 Hz frequency, 200 msn wavelenght, continuous symetrical biphasic current. Amptlitude was increased just below the motor range that cause flexion in toes.

Control group was followed with sham tibial nerve stimulation, which were performed by after starting electric current with TENS device, current were decreased and completely shut off. Sham stimulation was also applied for 6 weeks, 2 times in a week, 30 minutes.

After 6 weeks, both groups were evaluated with urodynamic study for the second time.

ICIQ-SF, King's Health Questionaire, Overactive Bladder Syndrome Symptom Scoring and urodynamic study parameters were examined in both pre- and post-treatment period.

Results were compared to see if there is any difference in the patients who followed with TNS and also pre-post treatment symptoms with PFTE and BT.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients who applied to our hospital with the illness interval of 6 months-24 months
* Cooperated patients with mini mental test 18 and above
* Patients who willing to be a participant
* Patients with scoring of OABSS 3 and above (at least 2 points must be gained from question 3.) will be evaluated with urodynamic study and only the patients with overactive detrusor findings during urodynamic study will be included.

Exclusion Criteria:

* Patients who not willing to be a participant
* Psychiatric or cognitive impairment, MMT < 18
* Spasticity that effects whole body, MAS 3 and above
* Urinary symptoms before stroke
* Global or sensorial aphasia
* Cardiac pacemaker
* Urinary tract infection
* Benign prostate hypertrophy
* Already receiving any treatment because of neurogenic bladder
* History of botulinum toxin injection to the detrusor muscle
* Active malignancy
* Pregnants
* Post-void residue above 200 mL

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Urodynamic Study Parameters | 6 weeks
  Maximum Cystometric Capacity (mL)
Overactive Bladder Symptom Scoring | 6 weeks
  A validated symptom scoring to detect the patients with overactive bladder symptoms and classifying them as low/moderate/high OABS. Higher results mean worse outcome

SECONDARY OUTCOMES:
ICIQ-SF | 6 weeks
  a subjective measure of severity of urinary loss and quality of life for those with urinary incontinence. Higher results mean worse outcome.
King's Health Questionaire | 6 weeks
  Subjective measure of severity of urinary incontinence consists of nine domains: two single-item domains (general health perceptions and incontinence impact), and seven multi-item domains (role limitations, physical limitations, social limitations, personal relationships, emotions, sleep/energy, and severity/coping. Higher results mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Umay Ekinci, MD, Principal Investigator — University of Health Sciences, Department of PM&R
Locations (1):
- Gaziler PMR, Training and Research Hospital, Department of PMR, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No